CLINICAL TRIAL: NCT07203079
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Comparing 48-Hour Post-Operative Administration of Oral Versus Intravenous Acetaminophen in Patients Undergoing Lumbar Spine Fusion Surgery
Brief Title: Oral Versus Intravenous Acetaminophen in Lumbar Spine Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Atman Desai, Professor of Neurosurgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 82641
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Acetaminophen 1000mg (Active Comparator): Participants take oral acetaminophen and placebo infusion for 48 hours within 2 hours after their spine surgery
  Interventions: Drug: Acetaminophen Oral Tablet; Drug: Placebo infusion
- Intravenous Acetaminophen 1000mg (Experimental): Participants take acetaminophen infusion and oral placebo for 48 hours within 2 hours after their spine surgery
  Interventions: Drug: placebo oral tablet; Drug: Acetaminophen infusion

INTERVENTIONS:
Drug: Acetaminophen Oral Tablet — Participants take 1000mg by mouth every 6 hours for a total of 8 doses (48 hours total) starting within 2 hours after their spine surgery.
  Other Names: Tylenol
  Arms: Oral Acetaminophen 1000mg
Drug: placebo oral tablet — Participants take one placebo tablet (matchable to tylenol) by mouth every 6 hours for a total of 8 doses (48 hours total) starting within 2 hours after their spine surgery.
  Arms: Intravenous Acetaminophen 1000mg
Drug: Acetaminophen infusion — Participants take 1000mg by intravenous infusion over 15 minutes every 6 hours for a total of 8 doses (48 hours total) starting within 2 hours after their spine surgery.
  Arms: Intravenous Acetaminophen 1000mg
Drug: Placebo infusion — Participants take 1000mg placebo by intravenous infusion over 15 minutes every 6 hours for a total of 8 doses (48 hours total) starting within 2 hours after their spine surgery.
  Arms: Oral Acetaminophen 1000mg

SUMMARY:
The goal of this study is to compare whether oral or intravenous acetaminophen works better for pain control in patients undergoing lumbar spine fusion surgery

ELIGIBILITY:
Inclusion Criteria:

* Plan for open lumbar laminectomy and fusion surgery (1-3 levels)
* Able to provide written informed consent
* Must be able to swallow pills

Exclusion Criteria:

* Medical contraindications to acetaminophen
* Emergency surgery
* Chronic pain unrelated to surgery
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) Pain Intensity Scale Score | postoperative time intervals: 2 hours (baseline), 6 hours, 12 hours, 24 hours, 36 hours, 48 hours
  Mean pain intensity scores post-operatively using 11-point Numerical Rating Scale (NRS) (scale ranges from 0 to 10, and higher score means higher pain)

SECONDARY OUTCOMES:
Length of Hospital Stay | After surgery until discharge, up to 10 days
Time to first ambulation after surgery | After surgery until discharge, up to 10 days
Quality of Life (EuroQol Questionaire) scale score | 48 hours, up to 1 month after surgery
  Participants rate their quality of life using the EuroQol-5D-5L questionnaire (scale from 1 to 5, 1 = no problem, 5 = severe problem)
Cumulative opioid consumption | After surgery until discharge, up to 10 days
  All opioid medications the patient takes after surgery will be converted to a morphine equivalent dose.
Healthcare cost during admission | After surgery until discharge, up to 10 days
  Cost of hospital stay obtained from participant's Electronic Medical Record
Number of participants with treatment-related hepatic toxicity | postoperative time intervals: 2 hours(baseline), 24 hours, 48 hours
  Values above the normal range for any of these four lab tests (AST, ALT, INR, bilirubin) will be considered hepatic toxicity
Number of participants with treatment-related skin rash | After surgery until discharge, up to 10 days, whichever is first
  Per clinician assessment
Change in Patient Global Assessment Scale Score | postoperative time intervals: 2 hours, 6 hours, 12 hours, 24 hours, 36 hours, 48 hours
  Participants report their overall wellbeing as measured by 5-point Likert scale (ranging from 0-5, where 1=very well; 2=well; 3=fair; 4=poor; and 5=very poor)
Time to first additional opioid medication dose | After surgery until discharge, up to 10 days
  Additional opioid pain medication as requested by the participant which is not scheduled
Total number of additional opioid medication doses | After surgery until discharge, up to 10 days
  Additional opioid pain medication as requested by the participant which is not scheduled

CONTACTS AND LOCATIONS:
Overall Officials: Atman Desai, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No